CLINICAL TRIAL: NCT00789581
Title: Phase III Study of Doxorubicin/Cyclophosphamide (AC) Followed by Ixabepilone vs. AC Followed by Paclitaxel in Patients With Triple-Negative Early-Stage Breast Cancer
Brief Title: A Randomized Trial of Ixempra Versus Taxol in Adjuvant Therapy of Triple Negative Breast Cancer
Acronym: TITAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 145; TITAN
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Adjuvant; Doxorubicin; Cyclophosphamide; Paclitaxel; Ixabepilone; TITAN
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; ixabepilone; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicin/cyclophosphamide, ixabepilone (Experimental): Doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 administered for 4 cycles of 21 days each, followed by ixabepilone at 40 mg/m2 given for 4 cycles of 21 days each.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Ixabepilone (Ixempra)
- Doxorubicin/cyclophosphamide, paclitaxel (Active Comparator): Doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 administered for 4 cycles of 21 days each, followed by paclitaxel at 80 mg/m2 weekly for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel (Taxol)

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 60 mg/m2
  Other Names: Adriamycin; hydroxydaunorubicin; Adriamycin PFS; Adriamycin RDF; Rubex
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cytophosphane
Drug: Ixabepilone (Ixempra) — Ixabepilone 40 mg/m2
  Other Names: Ixempra; azaepothilone B; BMS-247550
  Arms: Doxorubicin/cyclophosphamide, ixabepilone
Drug: Paclitaxel (Taxol) — Paclitaxel 80 mg/m2
  Other Names: Taxol
  Arms: Doxorubicin/cyclophosphamide, paclitaxel

SUMMARY:
This is a randomized, Phase III, open-label, multicenter study.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio to receive one of two different treatment arms. Patients in treatment arm 1 will receive AC followed by ixabepilone. Patients in treatment arm 2 will receive AC followed by weekly paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients greater than or equal to18 years of age.
2. Histologically confirmed invasive unilateral breast cancer (regardless of

   histology).
3. Early-stage breast cancer, defined as:

   * Node-positive disease: >0.2-mm metastasis in at least one lymph node (pN1mipN2b)OR
   * Node-negative, with primary tumor >1.0 cm (T1c-T3).
4. Definitive loco-regional surgery must have been completed as specified

   below:
   * Patients must have undergone either breast conservation surgery

     (i.e., lumpectomy) or total mastectomy.
   * Surgical margins of the resected section must be histologically free of

   invasive adenocarcinoma and ductal carcinoma in situ.
   * Surgical margins involved with lobular carcinoma in situ (LCIS) will not

   be considered as a positive margin; therefore, such patients will be eligible for this study without additional resection.
   * Patients must have completed axillary lymph node sampling for the pathologic evaluation of axillary lymph nodes as specified below:

   Sentinel node biopsy and/or either lymph node sampling procedure or axillary dissection.
5. Multicentric and multifocal invasive breast cancer is eligible if loco-regional surgery has been completed as described above.
6. Patients with synchronous bilateral cancers are eligible only if:

   * All cancers are of triple-negative phenotype, defined as ER-, PR-, HER2-.
   * Eligibility based on the highest stage grouping.
7. HER2 negative tumors. HER2 negativity must be confirmed by one of the

   following:
   * FISH-negative (FISH ratio <2.2), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.2).
8. Estrogen receptor negative (<10% staining by IHC for estrogen receptor).
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
10. Patient must be <= 84 days from having completed definitive primary breast surgery (either lumpectomy or mastectomy).
11. MammoSite brachytherapy radiation is acceptable if it is performed

    immediately following surgery and prior to chemotherapy. It is recommended that chemotherapy be started no earlier than 2 weeks following the removal of the MammoSite balloon catheter.
12. Adequate hematologic function, defined by:

    * Absolute neutrophil count (ANC) >1500/mm3
    * Platelet count >=100,000/mm3
    * Hemoglobin >9 g/dL
13. Adequate liver function, defined by:

    * AST and ALT <=2.5 x the upper limit of normal (ULN)
    * Total bilirubin <=1.5 x ULN (unless the patient has grade 1 bilirubin

    elevation due to Gilbert's disease or a similar syndrome involving slow

    conjugation of bilirubin).
14. Adequate renal function, defined by:

    * Serum creatinine <=1.5 x ULN
15. Complete staging work-up <=12 weeks prior to initiation of study treatment

    with computed tomography (CT) scans of the chest and abdomen/pelvis (abdomen/pelvis preferred; abdomen accepted), and either a positron emission tomography (PET) scan or a bone scan.
16. Adequate cardiac function, defined by a left ventricular ejection fraction

    (LVEF) value of >50% (or normal per institutional guidelines) by MUGA scan or echocardiogram (ECHO).
17. Adequate recovery from recent surgery. At least 1 week must have elapsed from the time of a minor surgery (i.e., sentinel node biopsy, port-acath (placement); at least 3 weeks must have elapsed from the time of a major surgery (i.e., lumpectomy, partial or total mastectomy, axillary lymph node dissection, breast reconstruction procedure).
18. Patients with previous history of invasive cancers (including breast cancer)

    are eligible if definitive treatment was completed more than 5 years prior to

    initiating current study treatment, and there is no evidence of recurrent disease.
19. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
20. Patient must be accessible for treatment and follow-up.
21. Women of childbearing potential must agree to use an acceptable method of birth control to avoid pregnancy for the duration of study treatment, and for 3 months thereafter.
22. All patients must be able to understand the investigational nature of the

study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. History of previous diagnosis of invasive breast cancer (unless treated >5 years previously with no recurrence). History of previously treated ductal carcinoma in situ (DCIS) is acceptable.
3. Any evidence or suspicion of metastatic disease other than ipsilateral

   axillary lymph nodes.
4. Any tumor >=T4 (cutaneous invasion, deep adherence, inflammatory breast cancer).
5. Previous anthracycline chemotherapy.
6. Concurrent use of CYP3A4 inhibitors from 72 hours prior to initiation of

   study treatment until the end of treatment with ixabepilone.
7. Previous treatment for this breast cancer (including neoadjuvant

   chemotherapy).
8. Previous cancer (with the exception of non-melanoma skin cancer or cervical carcinoma in situ) in the past 5 years (including invasive contralateral breast cancer).
9. Peripheral neuropathy of > grade 1 per NCI CTCAE v3.0.
10. Cardiac disease, including: congestive heart failure (CHF) > Class II per

    New York Heart Association (NYHA) classification; unstable angina (anginal symptoms at rest) or new-onset angina (i.e., began within the last 3 months), or myocardial infarction within the past 6 months; symptomatic CHF, unstable angina pectoris, cardiac arrhythmia, or cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
11. History of hypersensitivity to CremophorEL (polyoxyethylated castor oil) or

    a drug formulated in CremophorEL such as paclitaxel.
12. Use of any investigational agent within 30 days of administration of the first dose of study drug.
13. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
14. Concurrent severe, uncontrolled infection or intercurrent illness including,

    but not limited to, ongoing or active infection, or psychiatric illness/social

    situations that would limit compliance with study requirements.
15. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
16. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (70):
- United States (69):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Cancer Center of Huntsville, Huntsville, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - University of Southern Alabama, Mobile, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Wilshire Oncology Medical Group, La Verne, California
  - New Hope Cancer and Research Institute, Pomona, California
  - Eastern Connecticut Hematology Oncology, Norwich, Connecticut
  - Aventura Medical Center, Aventura, Florida
  - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Care, Davie, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Regional Cancer Center, Hollywood, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory/Winship Cancer Institute, Atlanta, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Medical College of Georgia Cancer Specialists, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Suburban Hem Onc, Lawrenceville, Georgia
  - Mid-Illinois Hematology & Oncology, Normal, Illinois
  - Hematology Oncology of the North Shore, Skokie, Illinois
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Kansas City Cancer Centers, Overland Park, Kansas
  - Cotton O'Neil Cancer Center, Topeka, Kansas
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mercy Hospital, Portland, Maine
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Fallon Clinic, Worcester, Massachusetts
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Fairview Medical Oncology Clinic, Edina, Minnesota
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Research Medical Center, Kansas City, Missouri
  - St. John's Clinic, Springfield, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - St. Clare's Hospital Oncology and Hematology, Denville, New Jersey
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Southern Oncology and Hematology, Vineland, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mid Ohio Oncology/Hematology, Inc./ The Mark H. Zangmeister Center, Columbus, Ohio
  - Hematology/Oncology Inc, Elyria, Ohio
  - Hickman Cancer Center (Flower Hospital), Sylvania, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Bux-Mont Oncology, Fox Chase Cancer Center, Rockledge, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Lowcountry Hematology Oncology, Mt. Pleasant, South Carolina
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Medical Oncology Methodist Hospital, Houston, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
- San Juan Hospital, San Juan, Puerto Rico

REFERENCES:
- [Background] Yardley DA, Arrowsmith ER, Daniel BR, Eakle J, Brufsky A, Drosick DR, Kudrik F, Bosserman LD, Keaton MR, Goble SA, Bubis JA, Priego VM, Pendergrass K, Manalo Y, Bury M, Gravenor DS, Rodriguez GI, Inhorn RC, Young RR, Harwin WN, Silver C, Hainsworth JD, Burris HA 3rd. TITAN: phase III study of doxorubicin/cyclophosphamide followed by ixabepilone or paclitaxel in early-stage triple-negative breast cancer. Breast Cancer Res Treat. 2017 Aug;164(3):649-658. doi: 10.1007/s10549-017-4285-6. Epub 2017 May 15. PMID 28508185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was designed to evaluate if doxorubicin+cyclophosphamide (AC) followed by ixabepilone was more effective than AC followed by standard weekly paclitaxel as adjuvant treatment for patients with operable triple negative breast cancer (TNBC). Between Dec 2008 and Jan 2011, 614 women with early-stage TNBC were enrolled from 63 U.S. sites.
Pre-assignment Details: Subjects were randomized in a 1:1 ratio to either of 2 arms: 306 to AC/Ixabepilone (Ixa); 308 to AC/paclitaxel (Pac). 489 patients completed all planned treatment with AC/Ixa or AC/Pac.
Groups:
- AC/Ixabepilone: Doxorubicin+cyclophosphamide (AC) every 3 weeks for 4 cycles (12 weeks), followed by ixabepilone every 3 weeks for 4 cycles (12 weeks).
  Doxorubicin: 60 mg/m2 Cyclophosphamide: 600 mg/m2 Ixabepilone (Ixempra): 40 mg/m2
- AC/Paclitaxel: Doxorubicin+cyclophosphamide (AC) every 3 weeks for 4 cycles (12 weeks), followed by weekly paclitaxel for 12 weeks.
  Doxorubicin: 60 mg/m2 Cyclophosphamide: 600 mg/m2 Paclitaxel (Taxol): 80 mg/m2
Period: AC Therapy
Arm/Group | AC/Ixabepilone | AC/Paclitaxel
Started (All randomized patients.) | 306 | 308
Completed (5 patients were randomized but never treated.) | 295 | 291
Not Completed | 11 | 17
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Disease recurrence | 3 | 1
Not completed — Intercurrent Illness | 1 | 0
Not completed — Never Treated | 1 | 4
Not completed — Other | 0 | 2
Period: Adjuvant Therapy
Arm/Group | AC/Ixabepilone | AC/Paclitaxel
Started | 295 | 291
Completed (4 patients completed AC therapy but did not initiate adjuvant treatment.) | 255 | 234
Not Completed | 40 | 57
Not completed — Never treated | 2 | 2
Not completed — Adverse Event | 20 | 44
Not completed — Withdrawal by Subject | 14 | 5
Not completed — Disease recurrence | 2 | 1
Not completed — Intercurrent Illness | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analyses of baseline characteristics, demographics and efficacy includes all randomized patients.
Groups:
- Ixabepilone: Doxorubicin and cyclophosphamide (AC) given every 3 weeks for 4 cycles, followed by ixabepilone every 3 weeks for 4 cycles.
  Doxorubicin: 60 mg/m2
  Cyclophosphamide: 600 mg/m2
  Ixabepilone (Ixempra): 40 mg/m2
- Paclitaxel: Doxorubicin and cyclophosphamide (AC) given every 3 weeks for 4 cycles, followed by paclitaxel weekly for 12 weeks.
  Doxorubicin: 60 mg/m2
  Cyclophosphamide: 600 mg/m2
  Paclitaxel (Taxol): 80 mg/m2
- Total: Total of all reporting groups
Arm/Group | Ixabepilone | Paclitaxel | Total
Number analyzed (Participants) | 306 | 308 | 614
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 124 | 93 | 217
  ≥50 years | 182 | 215 | 397
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 308 | 614
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 52 | 113
  White | 237 | 251 | 488
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 100 | 84 | 184
  Postmenopausal | 206 | 224 | 430

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: The percentage of participants with disease-free survival at 3 and 5 years. Disease-free survival (DFS) is measured from the time between randomization and the date of first documented disease recurrence, or death from any cause.
Time Frame: up to 5.25 years (63 months)
Population: The intent-to-treat population (all randomized patients) are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paclitaxel: Doxorubicin and cyclophosphamide (AC) given every 3 weeks for 4 cycles, followed by paclitaxel given weekly for 12 weeks.
  Doxorubicin: 60 mg/m2
  Cyclophosphamide: 600 mg/m2
  Paclitaxel (Taxol): 80 mg/m2
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 306 | 308
percentage of participants
  3-year DFS | 88.6 [84.3 to 91.8] | 88.8 [84.6 to 91.9]
  5-year DFS | 87.1 [82.6 to 90.5] | 84.7 [79.7 to 88.6]

2. Secondary Outcome: Overall Survival
Description: The percentage of participants with overall survival at 3 and 5 years are presented. Overall survival (OS) defined as the time between randomization to date of death from any cause.
Time Frame: up to 5.25 years (63 months)
Population: The intent-to-treat population (all randomized patients) are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 306 | 308
percentage of participants
  3-year OS | 92.4 [86.9 to 93.7] | 93.8 [90.2 to 96.1]
  5-year OS | 89.7 [85.5 to 92.7] | 89.6 [85.0 to 92.9]

ADVERSE EVENTS:
Time Frame: Every 3 weeks up to 28 weeks
Description: Adverse events (AEs) were collected for all patients who received at least 1 dose of treatment - from date of first treatment through the 30-day end of treatment period. All patients had at least one AE.
Arm/Group | Ixabepilone | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 58/305 | 50/304
Other Adverse Events (participants affected / at risk) | 305/305 | 304/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=305) | Paclitaxel (N=304)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 12 | 12
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 1
INFECTION (Infections and infestations) | 4 | 3
NAUSEA (Gastrointestinal disorders) | 3 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 1
SEPSIS (Infections and infestations) | 3 | 0
VOMITING (Gastrointestinal disorders) | 3 | 2
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
CELLULITIS (Infections and infestations) | 2 | 0
CHEST PAIN (General disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
NEUTROPHIL COUNT (Investigations) | 2 | 0
PAIN (General disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2
AORTIC STENOSIS (Vascular disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BREAST PAIN (Reproductive system and breast disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
CHEST WALL ABSCESS (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 3
DEPRESSION (Psychiatric disorders) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
FANCONI SYNDROME (Congenital, familial and genetic disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 3
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 2
SALPINGO-OOPHORECTOMY BILATERAL (Surgical and medical procedures) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0
ABSCESS LIMB (Infections and infestations) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 2
BREAST CELLULITIS (Infections and infestations) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
CATHETER SEPSIS (Infections and infestations) | 0 | 1
CATHETER THROMBOSIS (General disorders) | 0 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1
HAEMOGLOBIN (Investigations) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=305) | Paclitaxel (N=304)
Nausea (Gastrointestinal disorders) | 227 | 221 — All participants who had at least one dose of study drug.
Constipation (Gastrointestinal disorders) | 131 | 122 — All participants who had at least one dose of study drug.
Diarrhoea (Gastrointestinal disorders) | 112 | 114 — All participants who had at least one dose of study drug.
Vomiting (Gastrointestinal disorders) | 89 | 69 — All participants who had at least one dose of study drug.
Dyspepsia (Gastrointestinal disorders) | 53 | 51 — All participants who had at least one dose of study drug.
Stomatitis (Gastrointestinal disorders) | 52 | 51 — All participants who had at least one dose of study drug.
Gastroesophageal reflux (Gastrointestinal disorders) | 26 | 26 — All participants who had at least one dose of study drug.
Abdominal pain (Gastrointestinal disorders) | 20 | 22 — All participants who had at least one dose of study drug.
Fatigue (General disorders) | 250 | 251 — All participants who had at least one dose of study drug.
Mucosal Inflammation (General disorders) | 81 | 64 — All participants who had at least one dose of study drug.
Pyrexia (General disorders) | 47 | 50 — All participants who had at least one dose of study drug.
Oedema Peripheral (General disorders) | 36 | 58 — All participants who had at least one dose of study drug.
Pain (General disorders) | 47 | 27 — All participants who had at least one dose of study drug.
Alopecia (Skin and subcutaneous tissue disorders) | 214 | 208 — All participants who had at least one dose of study drug.
Rash (Skin and subcutaneous tissue disorders) | 33 | 47 — All participants who had at least one dose of study drug.
Nail disorder (Skin and subcutaneous tissue disorders) | 28 | 45 — All participants who had at least one dose of study drug.
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 19 — All participants who had at least one dose of study drug.
Pruritis (Skin and subcutaneous tissue disorders) | 18 | 16 — All participants who had at least one dose of study drug.
Neuropathy peripheral (Nervous system disorders) | 120 | 158 — All participants who had at least one dose of study drug.
Headache (Nervous system disorders) | 87 | 88 — All participants who had at least one dose of study drug.
Dysgeusia (Nervous system disorders) | 78 | 69 — All participants who had at least one dose of study drug.
Peripheral Sensory neuropathy (Nervous system disorders) | 55 | 65 — All participants who had at least one dose of study drug.
Dizziness (Nervous system disorders) | 37 | 41 — All participants who had at least one dose of study drug.
Paraesthesia (Nervous system disorders) | 16 | 19 — All participants who had at least one dose of study drug.
Arthralgia (Musculoskeletal and connective tissue disorders) | 106 | 87 — All participants who had at least one dose of study drug.
Bone Pain (Musculoskeletal and connective tissue disorders) | 83 | 46 — All participants who had at least one dose of study drug.
Myalgia (Musculoskeletal and connective tissue disorders) | 67 | 53 — All participants who had at least one dose of study drug.
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 47 | 40 — All participants who had at least one dose of study drug.
Back Pain (Musculoskeletal and connective tissue disorders) | 41 | 33 — All participants who had at least one dose of study drug.
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 37 | 22 — All participants who had at least one dose of study drug.
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 20 — All participants who had at least one dose of study drug.
Neutropenia (Blood and lymphatic system disorders) | 139 | 145 — All participants who had at least one dose of study drug.
Anaemia (Blood and lymphatic system disorders) | 104 | 119 — All participants who had at least one dose of study drug.
Leukopenia (Blood and lymphatic system disorders) | 69 | 83 — All participants who had at least one dose of study drug.
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 36 — All participants who had at least one dose of study drug.
Upper respiratory tract infection (Infections and infestations) | 34 | 20 — All participants who had at least one dose of study drug.
Urinary tract infection (Infections and infestations) | 26 | 28 — All participants who had at least one dose of study drug.
Sinusitis (Infections and infestations) | 21 | 33 — All participants who had at least one dose of study drug.
Cough (Respiratory, thoracic and mediastinal disorders) | 57 | 66 — All participants who had at least one dose of study drug.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 50 — All participants who had at least one dose of study drug.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 36 | 35 — All participants who had at least one dose of study drug.
Anorexia (Metabolism and nutrition disorders) | 56 | 43 — All participants who had at least one dose of study drug.
Dehydration (Metabolism and nutrition disorders) | 28 | 22 — All participants who had at least one dose of study drug.
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 28 — All participants who had at least one dose of study drug.
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 22 — All participants who had at least one dose of study drug.
Appetite decreased (Metabolism and nutrition disorders) | 19 | 18 — All participants who had at least one dose of study drug.
Insomnia (Psychiatric disorders) | 79 | 84 — All participants who had at least one dose of study drug.
Anxiety (Psychiatric disorders) | 27 | 40 — All participants who had at least one dose of study drug.
Depression (Psychiatric disorders) | 33 | 28 — All participants who had at least one dose of study drug.
hot flush (Vascular disorders) | 50 | 53 — All participants who had at least one dose of study drug.
Lacrimation increased (Eye disorders) | 24 | 26 — All participants who had at least one dose of study drug.
weight decreased (Investigations) | 22 | 16 — All participants who had at least one dose of study drug.
Neutrophil count (Investigations) | 21 | 13 — All participants who had at least one dose of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.